CLINICAL TRIAL: NCT03946865
Title: Reiki Therapy - an Intervention in Hematology/Oncology Cancer Patients Hospitalized in an Inpatient Setting - a Pilot Study.
Brief Title: Reiki Therapy - an Intervention in Hematology/Oncology Cancer Patients Hospitalized
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 restrictions and study personnel retirement
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-000456
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospitalized hematology/oncology cancer subjects (Experimental): Hospitalized hematology/oncology cancer will participate in Reiki Therapy
  Interventions: Other: Reiki Therapy

INTERVENTIONS:
Other: Reiki Therapy — Reiki is a healing practice that originated in Japan. Reiki practitioners place their hands lightly on or just above the person receiving treatment, with the goal of facilitating the person's own healing response.

SUMMARY:
Researchers are trying to determine if offering and providing reiki therapy in hospitalized hematology/oncology cancer subjects has any effects on symptoms and feeling during the subjects hospital stay.

DETAILED DESCRIPTION:
Primary Aim:

The primary aim of this study is to evaluate the feasibility of offering and providing Reiki Therapy in hospitalized hematology/oncology cancer patients. The intervention should not - interfere with the medical management of the participants. The investigators hypothesize that Reiki Sessions will be successfully integrated into conventional care of hospitalized cancer patients.

Secondary Aim:

The secondary aim is to evaluate the patient reported outcomes of their symptoms (pain, fatigue, anxiety) and feelings (happy, energetic, relaxed, and calm) before and after Reiki Therapy. The investigators' hypothesis is that there will be improvement of patients' symptoms/feelings score after the Reiki Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized hematology-oncology patients age 18 - 80
* Able to speak English and complete surveys
* Able to read, understand and sign inform consent.

Exclusion Criteria:

* Patient unwilling for reiki therapy.
* Unable to give written consent.
* Already having received or receiving other reiki treatment.
* Pregnant women. (As verbalized by participant)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in pain pain symptoms | Baseline, approximately 2 hours
  Measured using a numeric rating scale, where 0 is not at all and 10 is unbearable
Change in fatigue symptoms | Baseline, approximately 2 hours
  Measured using a numeric rating scale, where 0 is not at all and 10 is unbearable
Change in anxiety symptoms | Baseline, approximately 2 hours
  Measured using a numeric rating scale, where 0 is not at all and 10 is unbearable
Change in feeling happy | Baseline, approximately 2 hours
  Measured using a numeric rating scale, where 0 is best possible and 10 is worst possible
Change in feeling energized | Baseline, approximately 2 hours
  Measured using a numeric rating scale, where 0 is best possible and 10 is worst possible
Change in feeling relaxed | Baseline, approximately 2 hours
  Measured using a numeric rating scale, where 0 is best possible and 10 is worst possible
Change in feeling calm | Baseline, approximately 2 hours
  Measured using a numeric rating scale, where 0 is best possible and 10 is worst possible

CONTACTS AND LOCATIONS:
Overall Officials: Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials